CLINICAL TRIAL: NCT00311922
Title: Improving Care for Patients With Diabetes and Poor Numeracy Skills
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Vanderbilt University (Other)
Collaborators: Pfizer (Industry); Vanderbilt DRTC P&F Grant (DK20593) (Unknown); American Diabetes Association (Other)
Responsible Party: Russell Rothman, Vanderbilt University
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Health Services Research
Other Study IDs: IRB# 060128; DK20593 P&F 6 NIH/NIDDK
Record Dates: First submitted 2006-04-04; First posted 2006-04-06 (Estimated); Last update posted 2008-02-18 (Estimated); Status verified 2008-02

CONDITIONS: Diabetes
Keywords: Diabetes; Education; Health Literacy
MeSH Terms: conditions — Diabetes Mellitus | interventions — Control Groups

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Control (Active Comparator): Active Control Arm receives Comprehensive Diabetes Education
  Interventions: Behavioral: Control Group
- Intervention Arm (Experimental): Receives comprehensive education that is literacy/numeracy sensitive
  Interventions: Behavioral: Literacy/Numeracy oriented educational intervention

INTERVENTIONS:
Behavioral: Literacy/Numeracy oriented educational intervention — Comprehensive educational Intervention
  Arms: Intervention Arm
Behavioral: Control Group — Receives comprehensive education that is not literacy/numeracy sensitive
  Arms: Control

SUMMARY:
The aim of this research will be to perform a randomized controlled trial (RCT) of a new diabetes educational intervention that teaches self-management skills that compensate for poor numeracy skills among a sample of patients with diabetes and low numeracy.

DETAILED DESCRIPTION:
Results of the National Adult Literacy Survey (NALS) suggest that over 90 million adult Americans have poor quantitative skills. Numeracy, the ability to understand and use numbers and math skills in daily life, may be particularly important to patients with diabetes because caring for diabetes often requires self-management skills that rely on the daily application of math skills, such as counting carbohydrates, interpreting blood glucose monitoring, applying sliding scale insulin regimens, and calculating insulin to carbohydrate ratios. Presumably diabetes patients with poor numeracy have more difficulty with self-management and are at risk for poorer clinical outcomes, but to date, there are no published studies that rigorously examine the role of numeracy in diabetes. We have recently completed the initial development of a new scale to measure numeracy in patients with diabetes: the Diabetes Numeracy Test (DNT).

The aim of this research will be to perform a randomized controlled trial (RCT) of a new diabetes educational intervention that teaches self-management skills that compensate for poor numeracy skills among a sample of patients with diabetes and low numeracy. We hypothesize that a group of patients with poor numeracy who are taught self-management skills that accommodate their poor numeracy will have: (1) improved treatment satisfaction and perceived self-efficacy, (2) improved performance in self-management tasks, and (3) improved glycemic control compared to a control group that receives usual education.

ELIGIBILITY:
Inclusion Criteria:

1. Clinical diagnosis of Type 1 or 2 Diabetes;
2. most recent A1C greater than or equal to 7.0%;
3. Referred to the Diabetes Improvement Program for diabetes care;
4. Age 18-80;
5. English Speaking.

Exclusion Criteria:

1. Patients with corrected visual Acuity >20/50 using a Rosenbaum Pocket Vision Screener, or
2. Patients with a diagnosis of significant dementia, psychosis, or blindness.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 106 (Actual)
Dates: Start 2006-03; Primary Completion 2007-12 (Actual); Study Completion 2007-12 (Actual)

PRIMARY OUTCOMES:
A1C | 3 and 6 months

SECONDARY OUTCOMES:
Patient self-management behaviors | 3 and 6 months
Patient knowledge | 6 months
Patient satisfaction | 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Russell L Rothman, MD MPP, Principal Investigator — Vanderbilt University
Locations (1):
- Vanderbilt University Medical Center, Nashville, Tennessee, United States

REFERENCES:
- [Derived] Cavanaugh K, Wallston KA, Gebretsadik T, Shintani A, Huizinga MM, Davis D, Gregory RP, Malone R, Pignone M, DeWalt D, Elasy TA, Rothman RL. Addressing literacy and numeracy to improve diabetes care: two randomized controlled trials. Diabetes Care. 2009 Dec;32(12):2149-55. doi: 10.2337/dc09-0563. Epub 2009 Sep 9. PMID 19741187